CLINICAL TRIAL: NCT00005791
Title: Phase I Trial of Irinotecan, Cisplatin, and Fluorouracil in Patients With Advanced Solid Tumor Malignancies
Brief Title: Combination Chemotherapy in Treating Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067737; MSKCC-99065; NCI-G00-1743
Record Dates: First submitted 2000-06-02; First posted 2004-02-16 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2009-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Cisplatin; Fluorouracil; Irinotecan

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy in treating patients who have locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of weekly irinotecan in combination with weekly fluorouracil and cisplatin in patients with locally advanced or metastatic solid tumors. II. Determine the dose limiting toxicity for this combination regimen in this patient population. III. Establish a recommended phase II dose for this combination regimen in these patients. IV. Evaluate the safety and tolerability of this regimen in these patients. V. Observe any responses to this combination chemotherapy in these patients. VI. Measure in pretreatment biopsies levels of expression of thymidylate synthase, topoisomerase I, ERCC-1, thymidine phosphorylase, and dihydropyrimidine dehydrogenase as correlates to response or resistance to this combination chemotherapy in these patients.

OUTLINE: This is a dose escalation study of irinotecan and fluorouracil. Patients receive cisplatin IV over 30 minutes followed by fluorouracil IV over several minutes followed by irinotecan IV over 30 minutes on days 1, 8, 15, and 22. Treatment continues every 6 weeks in the absence of unacceptable toxicity or disease progression for a minimum of 3 courses. Cohorts of 3-6 patients receive escalating doses of irinotecan and fluorouracil until the maximum tolerated dose (MTD) of each is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicities. Patients are followed at 30 days and then until death.

PROJECTED ACCRUAL: A total of 3-36 patients will be accrued for this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed solid tumor malignancy not amenable to curative surgery or chemoradiation No CNS metastases, carcinomatous meningitis, or interstitial pulmonary fibrosis

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL AST no greater than 3 times upper limit of normal (ULN) (5 times ULN if liver metastases) No known Gilbert's disease Renal: Creatinine no greater than 1.5 mg/dL Calcium less than 12.0 mg/dL No symptomatic hypercalcemia Cardiovascular: No unstable angina No New York Heart Association class III or IV cardiac disease Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No active or uncontrolled infection No history of seizure disorder No uncontrolled diabetes mellitus, defined as random blood sugar 250 mg/dL or greater

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics No more than 1 prior chemotherapy regimen Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy and recovered No prior mantle irradiation, hemibody irradiation, or radiation to the pelvis or lumbar spine Surgery: See Disease Characteristics Other: No concurrent phenytoin, phenobarbital, or other antiepileptic medication No concurrent prochlorperazine on day of irinotecan administration No concurrent prophylactic loperamide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-10; Primary Completion 2002-07 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H. Ilson, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Ku GY, O'Reilly EM, Saltz LB, Schrag D, Maki RG, Kelsen DP, Ilson DH. Phase I study of weekly cisplatin, bolus fluorouracil and escalating doses of irinotecan in advanced solid tumors. Cancer Invest. 2009 May;27(4):402-6. doi: 10.1080/07357900802406327. PMID 19219674